CLINICAL TRIAL: NCT03445780
Title: Comparison of Distraction Methods for Pain Relief of Trigger Finger Injection
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No patients were enrolled; Senior author (Dr. Melamed) departed institution
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 17-01275
Record Dates: First submitted 2018-02-13; First posted 2018-02-26 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Trigger Finger
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- First Group (Experimental): Skin cooling with ethyl chloride spray will be used for 5 seconds prior to injection
  Interventions: Drug: Ethyl chloride spray
- Second Group (Experimental): The skin between the distal palmar crease and the palmo-digital crease and the palmo-digital crease will be pinched for 5 seconds prior to injection
  Interventions: Procedure: Pinching
- Third Group (Experimental): Skin cooling with ethyl chloride spray will be used for 5 seconds prior to injection as well as a second pinch to the skin between the distal palmar crease and the palmo digital crease
  Interventions: Drug: Ethyl chloride spray; Procedure: Pinching
- Fourth Group (Experimental): Subjects will sit behind a screen with a small opening large enough to introduce the injection hand. They will not see any of the procedure.
  Interventions: Procedure: No Site of Procedure

INTERVENTIONS:
Drug: Ethyl chloride spray — Skin cooling with ethyl chloride spray 5 seconds prior to injection
  Other Names: Bethamethasone
  Arms: First Group; Third Group
Procedure: Pinching — Skin between the distal palmar crease and the palmo digital crease will be pinched for 5 seconds prior to injection
  Arms: Second Group; Third Group
Procedure: No Site of Procedure — Subjects will sit behind a screen with a small opening large enough to introduce the injected hand. They will not see any of the procedure
  Arms: Fourth Group

SUMMARY:
The purpose of this study is to evaluate the best distraction mechanism during trigger finger injection in the outpatient setting. Temporary discomfort from the needle prick is highly feared by patients and is often accompanied by significant acute pain and distress during routine corticosteroid injection in the orthopedic outpatient setting. This study aims to examine 4 different distraction methods and their efficacy in reducing perceived pain, which will be evaluate using the VAS (visual analog pain score.) The three distraction methods will be ethyl chloride spray, adjacent pinch, ethyl chloride spray and pinch, and "screen" or looking away method.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Trigger Finger

Exclusion Criteria:

* Allergies to lidocaine, betamethasone, infection, pregnancy, 3 prior injection to the digit

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Analog Scale (VAS) Score | 1 Minute, 24 Hours
  A 10-cm scale will be shown to the patients, and they will be asked to choose the proper number, with 1 representing no pain and 10 symbolizing the most pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Eitan Melamed, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States